CLINICAL TRIAL: NCT04451213
Title: Magnetic Resonance Imaging and Neuro-Psychological Testing In Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19/MAR/7625
Record Dates: First submitted 2020-01-21; First posted 2020-06-30 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental)
  Interventions: Diagnostic Test: MRI head

INTERVENTIONS:
Diagnostic Test: MRI head — MRI head

SUMMARY:
CF is a complex, inherited illness that can affect many organs of the body. The investigators have found that some patients with CF have reported more problems with memory than would be expected at their age and that patients appear to be using memory strategies to overcome memory loss. The investigators intend to objectively test memory and examine MRI images of the brain of patients with CF.

DETAILED DESCRIPTION:
Patients with CF have several potential risk factors which may predispose them to memory problems. Because the CF population has historically only been young, this is not something that has been focused on. No research has currently identified whether patients with CF have a much earlier risk of developing cognitive impairment or how CF impacts on the brain.

There has not previously been work in this area of CF and the investigators are in a unique position with the Cardiff University Brain Research Imaging Centre (CUBRIC) and its expertise to be able to perform Magnetic Resonance Imagining (MRI) scans and neurocognitive testing on patients with CF for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged greater or equal to 30 years

  * A diagnosis of CF
  * Primary school education or above
  * Able to provide informed consent

Exclusion Criteria:

* Contraindications to MRI as found on the CUBRIC screening form (including presence of indwelling metal devices/clips)

  * Existing neurological disease affecting cognition (including stroke and traumatic brain injury)
  * Existing diagnosis of dementia documented in medical notes
  * Vascular complications of diabetes
  * Requiring supplemental oxygen -long term or overnight
  * Hepatic failure
  * Overt psychiatric disorders
  * Past or present alcohol or recreational drug misuse
  * Pregnancy
  * Current infection Smoker

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Objective memory scores | up to one year

SECONDARY OUTCOMES:
MRI head | up to one year
  the investigators will acquire structural and functional MRI data at 3T to explore brain health of CF patients compared to control data. Structural MRI will include T1 and T2 weighted anatomical images for group comparisons of brain morphology (volume, cortical thickness). T1 weighted images will also be used as reference images for all other MRI parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff and VAle University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No